CLINICAL TRIAL: NCT01796951
Title: Low Dose Aspirin Inhibition of COX-2 Derived PGE2 in Male Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Philip Lammers, Hematology/Oncology Clinical Fellow, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VR5137
Record Dates: First submitted 2013-02-14; First posted 2013-02-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Tobacco Use Disorder; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Aspirin; Celecoxib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Celecoxib, aspirin, followed by aspirin/celecoxib (Experimental): Celecoxib 200 mg twice daily x3 days, aspirin 325 mg daily x10 days, celecoxib 200 mb twice daily + aspirin 325 mg daily x 3 days
  Interventions: Drug: Aspirin 325 mg daily; Drug: Celecoxib 200 mg BID

INTERVENTIONS:
Drug: Aspirin 325 mg daily — In this single-arm trial, participants will take celecoxib 200 mg BID for 5 doses, followed by aspirin 325 mg daily for 10 days, followed by combination of celecoxib 200 mg BID for 5 doses and aspirin 325 mg daily for 3 days.
Drug: Celecoxib 200 mg BID — In this single-arm trial, participants will take celecoxib 200 mg BID for 5 doses, followed by aspirin 325 mg daily for 10 days, followed by combination of celecoxib 200 mg BID for 5 doses and aspirin 325 mg daily for 3 days.

SUMMARY:
Regular aspirin use has been associated with a reduction in the development of a number of different malignancies including lung cancer. The mechanism of aspirin's cancer prevention is not known. This study will evaluate whether once daily aspirin use can reduce the production of a protein named prostaglandin E2 (PGE-2), which is known to promote cancer. Specifically, this study will evaluate if aspirin can inhibit the production of PGE-2 by blocking an enzyme named cycloxygenase-2 (COX-2). To accomplish these goals, participants will take either aspirin 325 mg daily, celecoxib 200 mg twice daily, or the combination of both during various days of this 16-day study. Urine be collected to evaluate for PGE-2 production at 4 timepoints in this 16-day study.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age ≥35
* Current smoker of at least 10 cigarettes per day with history of ≥10 pack-years (py)
* Former smoker, quit no more than 15 years ago with a history of at least 25 py
* Ability to comply with the design of the study
* Capacity to freeze urine sample at participant's residence if this participant desires to store the urine specimens in this manner
* Baseline urine PGE-M > 13 ng/mg creatinine
* Serum thromboxane > 150 μg/L

Exclusion Criteria:

* History of aspirin use 1-14 days prior to screening
* NSAID (ibuprofen, naprosyn, meloxicam, etc) use 1-7 days prior to screening
* Inhaled glucocorticoid use 1-7 days prior to screening
* Systemic glucocorticoid use 1-14 days prior to screening
* History of peptic ulcer disease
* Current or recent clinically significant bleeding
* Allergy, intolerance or contraindication to aspirin or NSAID use
* Thrombocytopenia (platelet count < 100,000) in 30 days prior to screening visit
* Severe hepatic insufficiency
* GFR < 30 mL/min/1.73 m2 in 30 days prior to screening visit
* History of aspirin or celecoxib allergy
* Elevated INR (>1.5) in 30 days prior to screening visit
* Current diagnosis of malignancy or history of non-skin malignancy in last 5 years
* Current use of systemic anticoagulants (e.g., warfarin (Coumadin), enoxaparin (Lovenox), Fondaparinux (Arixtra), dabigatran (Pradaxa))
* Diagnosis of COPD
* Intake of > 250 mg of fish oil supplementation daily

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in COX-2 dependent urinary PGE-M (ng/mg Cr) production after 16 days of aspirin treatment | 16 days
  Baseline urinary PGE-2 metabolite (PGE-M) will be measured. Then after 3 days of COX-2 blockade with celecoxib, it will again be measured. Participants will then undergo 10 days of treatment with aspirin and urinary PGE-M will be measured. Finally, participants will be treated with combined aspirin and celecoxib for 3 days and urinary PGE-M will be measured one last time. Using these values, the degree of aspirin inhibition of COX-2 specific urinary PGE-M production can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: John A Oates, MD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States